CLINICAL TRIAL: NCT04999085
Title: Geriatric-assessment-guided Interventions to Address Functional Deficits in Older Adults Undergoing Treatment for Multiple Myeloma
Brief Title: Geriatric-assessment Interventions to Address Functional Deficits in Older Adults w Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC 2101; 2021YIA-7316118933 (Other Grant/Funding Number: Conquer Cancer Foundation)
Record Dates: First submitted 2021-08-02; First posted 2021-08-10 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma; Myeloma; Disability Physical; Disabilities Multiple
Keywords: Geriatric assessment; Supportive care; Disability; Functional assessment
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Single-arm pilot study of supportive care interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Experimental)
  Interventions: Other: Supportive care interventions

INTERVENTIONS:
Other: Supportive care interventions — Subjects will be referred to specialists and/or supportive care interventions based on issues/deficits identified on a baseline geriatric assessment. These interventions will be selected based on deficits or problems identified on baseline assessments. These include referral to physical/occupational therapy for those with physical deficits (Activities of Daily Living impairment, Instrumental Activities of Daily Living impairment, Timed Up and Go, or falls), to optometry/ophthalmology (for visual impairment), to audiology (for hearing impairment), to pharmacist (for polypharmacy), and to cancer center support program (for Mental Health Index 13 criteria).

SUMMARY:
Myeloma is the second most common type of blood cancer in the United States. Myeloma most commonly affects older adults. While some younger individuals do get myeloma, the average age when people are first diagnosed with myeloma is around 69 to 70.

Along with having a higher risk for myeloma, older adults have an increased chance of developing other health problems or issues. However, not everyone ages in the same way. Some older adults experience major changes in health or degree of independence at relatively younger ages, while others remain quite healthy for many years. The specific issues that develop with age can also vary from person to person. One older adult may face difficulties with vision or hearing, while another may develop memory problems.

Historically, cancer doctors have not done a very good job identifying these non-cancer issues. As a result, research has focused on better ways to systematically pick up on issues that may impact cancer outcomes or quality of life. The outgrowth of this research is assessments and questionnaires referred to as "comprehensive geriatric assessments," which evaluate the health and functionality of older adults thoroughly but efficiently. In both myeloma and other types of cancer, problems identified through geriatric assessments have been shown to predict how likely people are to develop side effects of cancer treatment and predict how long people are likely to live with cancer.

Prior research has not addressed how best to help with the issues picked up through a geriatric assessment among patients undergoing treatment for myeloma, although a number of effective interventions have been shown to benefit older adults with similar problems in other settings. Therefore, the current study will test a strategy of systematically screening older adults undergoing myeloma treatment for geriatric-assessment-related deficits and referring participants to appropriate services and resources. The geriatric assessment in this study includes tests of mobility, memory, vision, hearing, and nutrition as well as questions about symptoms and social support. Individuals who have deficits in one of these areas will be referred to relevant services and resources such as physical therapy, a pharmacist, or the cancer center support program. They will then repeat the same assessment three months later, and the results will be compared to their original assessment to see if the deficit has improved, with particular attention to mobility and social support.

DETAILED DESCRIPTION:
STUDY OUTLINE

Study participants complete a baseline Geriatric Assessment and European Organization for Research and Treatment of Cancer (EORTC) Quality of Life of Cancer Patients (QLQ) Core 30 (C30) and Myeloma supplement (MY20) questionnaires, either at the time of enrollment or as part of previous research studies.

Based on these assessments, an intervention strategy is developed by Study Team. These interventions largely consist of referrals to relevant specialists and existing services. These recommendations are communicated to the study participant, and participant-approved intervention referrals are made.

Following an initial appointment with these specialists, further follow-up will be determined based on the subject and specialist without input from the Study Team.

At three months from enrollment, study participants will be asked to complete a follow-up geriatric assessment, repeat EORTC questionnaires, and a satisfaction /feedback survey.

Duration of Therapy:

For patients referred to specialists as above, the duration of treatment or care with the specialist will be determined based on an agreement between the specialist and study participant.

Duration of Follow-up:

As part of this study, participants will only be followed through the three-month follow-up assessment described above. For subjects participating in or recruited from other research studies, follow-up according to those other protocols will continue.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 60 years or older with a confirmed diagnosis of multiple myeloma currently undergoing or planned to begin treatment for multiple myeloma.
* Enrollment in an existing registry of individuals with plasma cell disorder (ClinicalTrials.gov identifier NCT03717844; institutional protocol # LCCC1728)
* Be willing and capable of providing informed consent.

Presence of at least one intervenable deficit on the most recent registry assessment:

* Activities of daily living score < 14.
* Instrumental activities of living score < 14.
* Timed Up and Go test = 14 seconds (or unable to complete the test).
* One fall in the prior 6 months.
* Eyesight poor or worse.
* Hearing poor or worse.
* Number of daily medications 10 or greater.
* Mental Health Index-13 Depression score 12 or greater.
* Mental Health Index-13 Anxiety score 6 or greater.

Exclusion Criteria:

* Has dementia, altered mental status, or any psychiatric or co-morbid condition prohibiting the understanding or rendering of informed consent.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Jensen, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The N.C. Cancer Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina (UNC) Lineberger Comprehensive Cancer Center — http://unclineberger.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 11/15/2021 through 05/04/2023 at one cancer center in North Carolina. Subjects were enrolled in the study between 12/01/2021 - 12/15/2022.
Pre-assignment Details: Subjects were enrolled in the study between 12/01/2021- 12/15/2022, at one cancer center in the United States. A total of 16 participants consented, were found eligible, and started to study.
Period: Overall Study
Arm/Group | Supportive Care
Started | 16
Completed | 15
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: A total of 16 participants consented, were found eligible, and started to study. between 12/01/2021- 12/15/2022.
Arm/Group | Supportive Care
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 75.69 [66 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Intervention Attendance (Feasibility)
Description: Attendance at at least one appointment for a specialty / supportive care resource to which the subject is referred. The result is reported as the number of participants who attend at least one such appointment.
Time Frame: Up to 3 months from enrollment
Population: Subjects who started the study completed at least one study intervention.
Measure: Number; unit: percentage of participants
Arm/Group | Supportive Care
Number analyzed (Participants) | 16
percentage of participants | 50

2. Secondary Outcome: Subject Satisfaction With Program (Acceptability)
Description: Subject satisfaction with the intervention program, will be assessed by a single-item 5-point from 1 to 5, Likert scale response, with higher scores indicating greater satisfaction and lower scores indicating less satisfaction. The mean score reported by study participants will be reported.
Time Frame: 3 months from enrollment
Population: Subjects who started the study completed study interventions and followed up 3 months.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Supportive Care
Number analyzed (Participants) | 15
score on a scale | 4.4 [3.7 to 5]

ADVERSE EVENTS:
Time Frame: Up to 3 months. The protocol does not require adverse event assessment.
Description: The protocol does not require adverse event assessment. Adverse Event Data was not collected.
Arm/Group | Supportive Care
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT04999085/Prot_SAP_000.pdf